CLINICAL TRIAL: NCT01756001
Title: Using Behavioral Economics to Promote Medication Adherence and Habit Formation
Brief Title: GlowCaps Adherence Randomized Control Trial
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Harvard University (Other); National Bureau of Economic Research, Inc. (Other); Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 816493; 10035604 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2012-12-06; First posted 2012-12-24 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Medical Adherence
MeSH Terms: interventions — Compensation and Redress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control Arm: Arm 1 will be the Control arm, in which subjects will be instructed to use the GlowCap for their chronic disease medication but will not be provided with any specific incentive for taking the medication or with any aid in remembering to do so.
  Interventions: Device: GlowCap
- Reminder Arm: Arm 2 will be the Reminder arm with daily email, text message, or phone call reminders for intervention. Subjects will be told that to aid in daily adherence to the medication, they will be provided with reminders for the first three months of the study and possibly again later in the study. At the start of the study, subjects will be given the option to receive daily email reminders, text message reminders, or daily (automated) phone call reminders to take their pill, each at a time of day that they choose. The default setting will be for subjects to receive both text and email reminders at 8AM each day. Subjects will be instructed on how to change their settings if they would like to receive a different set of reminders at different points in time.
  Interventions: Device: GlowCap; Behavioral: Daily email, text message, or phone call reminders
- Incentives Arm: Arm 3 will be the financial incentives arm, in which subjects will be paid for adherence. Their total earnings will be administered at the end of the experiment through the WTH platform.
  Interventions: Device: GlowCap; Behavioral: Paid for adherence
- Incentives and Reminders Arm: Arm 4 will be the financial incentives and reminders arm, in which subjects will be paid for adherence. Their total earnings will be administered at the end of the experiment through the WTH platform. They will also receive daily email, text message, or phone call reminders for intervention. Subjects will be told that to aid in daily adherence to the medication, they will be provided with reminders for the first three months of the study and possibly again later in the study. At the start of the study, subjects will be given the option to receive daily email reminders, text message reminders, or daily (automated) phone call reminders to take their pill, each at a time of day that they choose. The default setting will be for subjects to receive both text and email reminders at 8AM each day. Subjects will be instructed on how to change their settings if they would like to receive a different set of reminders at different points in time.
  Interventions: Device: GlowCap; Behavioral: Daily email, text message, or phone call reminders; Behavioral: Paid for adherence

INTERVENTIONS:
Device: GlowCap — The main research instrument is an electronic pill bottle called GlowCaps (by Vitality) that has the ability to transmit adherence data to the Way to Health (WTH) web portal. The investigators will measure adherence by counting the number of properly taken doses during the final four weeks of the study. Each time the pill bottle is opened, a date- and time-stamped wireless signal is sent to the Vitality server via the AT&T cellular network which will then be uploaded to the Way to Health portal for aggregation.
Behavioral: Daily email, text message, or phone call reminders
  Groups: Incentives and Reminders Arm; Reminder Arm
Behavioral: Paid for adherence
  Groups: Incentives Arm; Incentives and Reminders Arm

SUMMARY:
This randomized control trial will explore interventions to promote medication adherence using a novel electronic device that can track daily pill use. 500 subjects will be randomized into 4 arms of the experiment. In addition to a control arm, our three arms will be: reminders, financial incentives, and reminders and financial incentives.

DETAILED DESCRIPTION:
The investigators aim to study simple "behavioral economics" interventions that rely on consumer engagement to overcome cognitive and motivational barriers to medication adherence. Our goals are threefold: (1) to analyze which interventions are most effective in promoting medication adherence; (2) to analyze which interventions are most effective in promoting long-term habits that persist even when the interventions are removed; and (3) to understand how various patient characteristics (e.g. age or risk preferences) predict adherence or treatment receptivity. The investigators plan to track daily adherence of patients to a prescribed chronic disease drug using a new technology that electronically monitors when a pill bottle has been opened. In our control condition, patients will be monitored but not be provided with any reminders, adherence information, or incentive to adhere to their medication. Our three additional treatments will be either: (1) provide the patient with a daily email, text message, or phone call reminder to take the pill; (2) pay patients for each day that they take their pill (3) provide the patient with a daily email, text message, or phone call reminder to take the pill and pay patients for each day that they take their pill.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with chronic disease
* age 18-84

Exclusion Criteria:

* all patients not meeting inclusion criteria
* people who report that they currently use a day-of-the-week pill bottle
* people for whom AT&T does not have reliable wireless service for the Glowcap to communicate with the Way To Health platform

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 to 64, receiving coverage from Independence Blue Cross (IBX), and receiving an oral prescription for chronic disease. Subjects were recruited from a base pool of eligible subjects identified by IBX as patients who have been identified as having the lowest medication possession ratios.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Number of doses taken | 40 weeks
  This is a randomized controlled study with 5 arms - 1 control and 4 interventional. The primary outcome will be the number of doses taken as directed during the course of the study.

SECONDARY OUTCOMES:
Subjects' reported wellbeing | 13 weeks
  Secondary outcomes will be subjects' reported wellbeing and subjects' evaluations of the various interventions. Secondary outcomes will also include claims and cost of care for subjects from Blue Cross Blue Shield (BCBS) of Massachusetts for two years after the intervention.
Subjects' evaluation of the various interventions | 26 weeks
  Secondary outcomes will be subjects' reported wellbeing and subjects' evaluations of the various interventions. Secondary outcomes will also include claims and cost of care for subjects from Blue Cross Blue Shield (BCBS) of Massachusetts for two years after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Judd Kessler, Principal Investigator — University of Pennsylvania; Dmitry Taubinsky, Principal Investigator — Harvard University; Eric Zwick, Principal Investigator — Harvard University
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers. All data will be de-identified, aggregated, and summarized.

REFERENCES:
- [Background] Acland, D and Levy, M. Habit Formation and Naivete in Gym Attendance: Evidence from a Field Experiment. Mimeo 2010.
- [Background] Allcott H. Social norms and energy conservation. Journal of Public Economics 2011; 95: 1982-1095.
- [Background] Cutler DM, Everett W. Thinking outside the pillbox--medication adherence as a priority for health care reform. N Engl J Med. 2010 Apr 29;362(17):1553-5. doi: 10.1056/NEJMp1002305. Epub 2010 Apr 7. No abstract available. PMID 20375400
- [Background] Deci, E. Effects of externally mediated rewards on intrinsic motivation. Journal of Personality and Social Psychology 1971; 18: 105-115.
- [Background] Doshi JA, Zhu J, Lee BY, Kimmel SE, Volpp KG. Impact of a prescription copayment increase on lipid-lowering medication adherence in veterans. Circulation. 2009 Jan 27;119(3):390-7. doi: 10.1161/CIRCULATIONAHA.108.783944. Epub 2009 Jan 12. PMID 19139387
- [Background] Gerber AS, Green DP, Larimer CW. Social pressure and voter turnout: evidence from a large- scale field experiment 2008; 102:22-48.
- [Background] Gneezy U, Rustichini A. Pay enough or don't pay at all. Quarterly Journal of Economics 2000; 115: 791-810.
- [Background] Gneezy U, Rustichini A. A fine is a price. Journal of legal studies 2000; 29: 1-18.
- [Background] Karlan D, McConnell M, Mullainathan S, Zinman J. Getting to the top of mind: How reminders increase saving. Mimeo 2010.
- [Background] Long JA, Helweg-Larsen M, Volpp KG. Patient opinions regarding 'pay for performance for patients'. J Gen Intern Med. 2008 Oct;23(10):1647-52. doi: 10.1007/s11606-008-0739-1. Epub 2008 Jul 29. PMID 18663540
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Schultz PW, Nolan JM, Cialdini RB, Goldstein NJ, Griskevicius V. The constructive, destructive, and reconstructive power of social norms. Psychol Sci. 2007 May;18(5):429-34. doi: 10.1111/j.1467-9280.2007.01917.x. PMID 17576283
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784